CLINICAL TRIAL: NCT04039880
Title: An Open-Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Olorofim Administered Via the Oral Route to Healthy Male Subjects
Brief Title: Absorption, Metabolism and Excretion of 14C-olorofim in Man
Acronym: hAME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: F901318-01-09
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-08

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections | interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (mass balance) (Experimental): evaluation of mass balance and metabolite profiling
  Interventions: Drug: Olorofim
- Cohort B (biliary evaluation) (Experimental): evaluation of biliary elimination
  Interventions: Drug: Olorofim

INTERVENTIONS:
Drug: Olorofim — single oral dose (120 mg, 3.7 MBq)
  Other Names: F901318

SUMMARY:
Single-centre, open-label, non-randomised, single dose study in 2 cohorts of healthy subjects. It is planned to enrol 6 healthy male subjects in Cohort A (standard mass balance and metabolite profiling cohort) and up to 6 subjects in Cohort B (biliary evaluation cohort); each subject will receive a single oral administration of 120 mg [14C]-olorofim oral solution containing approximately 3.7 MBq (100 µCi).

DETAILED DESCRIPTION:
Subjects will be screened up to 28 days prior to dosing and eligible subjects will be admitted to the Clinical Research Unit (CRU) on the day prior to dosing (Day-1). Each subject will be dosed on the morning of Day 1 after an overnight fast.

Cohort A:

Subjects will remain resident in the CRU up to 336 h post-dose (Day 15), with whole blood, plasma, urine and faeces collected throughout this period. There may be up to two further 24 h residency periods (Days 21 to 22 and Days 28 to 29) for collection of plasma, urine and faeces if discharge criteria are not met.

Cohorts B1 and B2:

Subjects will remain resident in the CRU up to 96 h post-dose (Day 5) for collection of plasma, urine, faeces and bile. Subjects will return for a short follow-up visit on Day 10. Cohort B1 subjects will have bile sampling up to 6 h postdose and Cohort B2 subjects will have bile sampling up to 12 h postdose. Cohort B divided into 2 sub-cohorts for logistical reasons only.

ELIGIBILITY:
Inclusion Criteria:

* healthy males age 18 to 55 years of age with body mass index of 18 to 30 kg/m2 (inclusive), and a body weight of 50 to 100 kg (inclusive).
* Subjects must be in good health as determined by a medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is NOT acceptable).
* Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day).

Exclusion Criteria:

* Subjects with or history of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatry, respiratory, metabolic, endocrine, ocular haematological or other major disorders as determined by the investigator
* Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration
* Current smokers and those who have smoked or used nicotine containing products (eg electronic cigarettes) within the 3 months prior to check-in.
* Radiation exposure, including that from the present study exceeding 1 mSv in the last 12 months or 5 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mass balance | 28 days
  % dose recovered in urine and faeces
Metabolite profiling | 15 days
  number of metabolites in plasma, urine and faeces > 10% of circulating radioactivity

SECONDARY OUTCOMES:
biliary elimination | 5 days
  radioactivity present in bile (ug equiv/g)
Maximum plasma concentration (Cmax) for olorofim, F902412 and total radioactivity | 15 days
time of maximum plasma concentration (Tmax) for olorofim, F902412 and total radioactivity | 15 days
elimination half life (t1/2) for olorofim, F902412 and total radioactivity | 15 days
Area under plasma concentration curve (AUC) for olorofim, F902412 and total radioactivity | 15 days
Number of subjects with treatment-related adverse events | 28 days
Number of subjects with clinically significant change from baseline in vital signs, laboratory parameters, and electrocardiogram findings | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jaap van Lier, MD, Principal Investigator — PRA
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No